CLINICAL TRIAL: NCT07373093
Title: Predictors of Measles Vaccine Hesitancy in New York State
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: WOLL-MEASLES-01
Record Dates: First submitted 2025-12-30; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Measles Vaccination
Keywords: measles; pediatric emergency department
MeSH Terms: conditions — Measles | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — The study population included caregivers of children aged 1-6 years old presenting to the emergency department during the study period. Convenience sampling was used to identify eligible participants. Survey was administered.

SUMMARY:
Under-immunization rates for childhood immunizations in the United States range from 8-20%. Previous studies have demonstrated that pediatric patients are most likely to be under-immunized for seasonal immunizations. The aim of this study is to explore the factors and facilitators contributing to measles immunization hesitancy. A secondary aim is to explore the impact of hypothetical contexts on measles immunization hesitancy. The results of this study may identify potential disparities in measles immunization coverage and potential solutions for addressing those disparities.

DETAILED DESCRIPTION:
SUBJECT POPULATION (WHO, WHAT, WHERE)

Aim 1: Guardians of patients 1 year to 6 years old presenting to the pediatric emergency department between 6/1/2025 and 6/1/2026 will be eligible. It is expected that approximately 800 parental encounters will be enrolled at AMC. Parents of children meeting the above inclusion and exclusion criteria will be approached for consent to participate in the study by convenience sampling weekdays 0900-1700. All consenting guardians will complete a brief survey to assess parental demographics and child immunization history. All participants who identify that a child is under-immunized for measles (i.e., did not receive 1st MMR immunization at 1 year of age OR 2nd MMR immunization at 4 years of age) will go on to complete a comprehensive survey to assess immunization beliefs.

Aim 2: In a private location, research assistants (RA) will randomly sample patients between 1 and 6 years of age in the pediatric ED and approach the patient's caregivers for participation in the survey if eligible. Caregivers will give written consent to participate in the survey. Caregivers will complete the survey in the ED on a private tablet. All guardians who complete the comprehensive survey will be randomized to receive one of four patient-centered immunization messages. The guardian will then be asked again if there is intent to immunize the child against RSV this season and if acceptance of immunization would occur if administered at the current visit.

Patient Sampling The RA will screen patients using convenience sampling methodology.

Patient recruitment, enrollment, and progress through the study Once a patient is screened and determined to be eligible, the RA will review the patient's ED electronic health record (dashboard or face sheet) and record (in a REDCap database) the following de-identified information: race/ethnicity, gender, ESI level, insurance status, and chief complaints. [Please see data collection form/survey for further details collected.]

Collecting de-identified data from patient charts poses no or minimal risk to the patient and is generally considered acceptable without prior patient consent. This information will be retained for all patients, even if participation in the survey portion is refused, as the information is helpful to understand which patients refused participation and which patients participated in the study to comment on potential sampling bias. These demographic data are (a) de-identified, (b) readily available, (c) able to be collected as a chart review without individual patient consent, (d) not sensitive information, and (e) for patients who do not wish to participate in the survey, not linked in any way with the study questions. The information collected allows the investigators to compare the demographics of participants and non-participants and therefore ensure that the sample is not biased.

If a patient meets the inclusion criteria, an RA will administer the consent for collection of the patient's name, medical record number, and survey responses.

D. DATA ANALYSIS The following data will be collected: Age, Gender, Race, Ethnicity, State of residence, parental age, parental education level, household income, insurance status, parental report of immunization status, and the reason for under-immunization if applicable. The sub-investigators will perform the data analysis at Albany Medical Center (AMC) using an AMC-approved password-protected PC. Storage of files will be on a password-protected departmental drive. A password-protected master key document will be used to store identifiers separately from other study variables, which will be collected and stored through REDCap.

The primary outcome is the demographic variables and immunization beliefs associated with RSV under-immunization. Survey responses will be used to stratify outcomes according to child age, Gender, Race, Ethnicity, State of residence, parental age, parental education level, household income, insurance status, and sources of health information. The secondary outcome is improvement in immunization confidence (defined as converting from "definitely not intent, unsure about intent, or probably not intent" to "intent") stratified by patient-centered immunization messaging.

Sample Size Considerations Approximately 800 patients are planned for enrollment at AMC.

E. RISKS The primary risk to individuals whose data are being used in this study is the potential breach of confidentiality of research data. Confidentiality is recognized as of foremost importance, and a series of standard practices will be used to protect the confidentiality of study participants. The risk of loss of confidentiality is considered a high priority in any project, and effective safeguards are in place to assure that confidentiality is not breached in the proposed project.

F. BENEFITS This research project aims to better understand patient risk for vaccine-preventable infections. All patients stand to benefit from advances in health care quality, safety, and efficiency. Risks to study subjects are believed to be minimal. The projected increase in the value of health care is exponentially higher than the investment.

The project will enable:

1. Standardized communication of vital history elements
2. Electronic surveillance
3. Error prevention
4. Reporting of quality metrics, cost, and outcomes

G. CONFIDENTIALITY Only project personnel directly involved in the study will have access to identified patient data and medical charts at the respective site. All project personnel with access to patient data will be trained in the proper handling of such data. Each study subject will be assigned a unique study identification number linked to the medical record number. Existing procedures will be used to ensure that individual patient identifiers are kept separate from analysis files and are available to project personnel on a need-to-know basis. PHI linked (patient name and MR number) to the study number will be kept in a separate password-protected Excel file from the remaining data points. This file will be stored on a secure AMC server with user-permission access. This master key will be destroyed once data collection is closed and the adjudication process completed for enrolled subjects. Data collection forms not including PHI will be recorded in REDCap on a secure AMC server. This de-identified data set will remain following completion of subject enrollment and adjudication. The data will be analyzed by Dr. Ashar Ata (AMC biostatistician).

H. OPTIONS Parents of patients may refuse participation without impact on care provided in the ED.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* -The patient is critically ill- Any life-threatening condition that requires pharmacological and/or mechanical support of vital organ functions, i.e. shock, moderate to severe asthma exacerbation, airway obstruction, anaphylaxis, etc.
* The patient presents with major (i.e. leveled) trauma
* The patient presents with concern for physical or sexual assault
* The patient presents with need for child protective service evaluation
* The patient or guardian are not English speaking
* The patient presents in custody of a juvenile detention center or law enforcement
* The patient presents without a consenting parent or legal guardian present at time of evaluation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of patients aged 1 year up to and including 6 years of age who present to the AMC pediatric ED between 7/1/2025 and 8/4/2025
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Caregiver Measles Vaccination Intent | Baseline (during pediatric emergency department visit)
  Caregiver intent to vaccinate their child against measles, measured using a single survey item with categorical responses ("yes," "unsure," "probably not," or "definitely not") and reported as the proportion of caregivers classified as intent ("yes") versus non-intent ("unsure," "probably not," or "definitely not") at baseline.

SECONDARY OUTCOMES:
Change in Caregiver Measles Vaccination Intent After Message Exposure | Immediately after provider message exposure during the same emergency department visit
  Change in caregiver measles vaccination intent following exposure to a standardized provider message, measured as the proportion of initially non-intent caregivers who changed classification from non-intent to intent after receiving one of four terminology-based messages ("vaccine," "immunization," "shot," or "medicine").

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol: Measles immunization (2026-01-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT07373093/Prot_000.pdf